CLINICAL TRIAL: NCT02801058
Title: Ultrasound Evaluation of Changes in Diaphragmatic Motion and Contractility Induced by Osteopathic Manipulative Techniques: a Prospective, Randomized, Double Blinded, Case vs Sham vs Control Clinical Trial.
Brief Title: Ultrasound Evaluation of Changes in Diaphragm Induced by Osteopathic Manipulative Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scarlata, Simone, M.D. (Other)
Responsible Party: Principal Investigator, Simone Scarlata, Scarlata, Simone, M.D., Scarlata, Simone, M.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SS-2016-1
Record Dates: First submitted 2016-06-09; First posted 2016-06-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Diaphragm; Respiratory Muscles; Osteopathic Medicine; Ultrasonography
Keywords: Osteopathic manipulative treatment; Abdominal Diaphragm mobility; Thoracic Ultrasounds
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Simple observation
- Shame (Sham Comparator): Light touch manipulative simulation
  Interventions: Other: Osteopathic manipulative treatment
- Treatment (Experimental): Osteopathic manipulative techniques on the abdominal diaphragm
  Interventions: Other: Osteopathic manipulative treatment

INTERVENTIONS:
Other: Osteopathic manipulative treatment — Osteopathic manipulative techniques on thoracic diaphragm
  Arms: Shame; Treatment

SUMMARY:
A wide number of osteopathic techniques focusing on diaphragm have been proposed but, although systematically and efficiently used, there is a general lack of evidences able to clarify how and to which extent osteopathic manipulative treatment (OMT) on diaphragm is effective and determines a modification in muscles contractility and motion as well as an objective determination of the benefit on the patients receiving treatment.

This study therefore aims at investigating whether, and how, a single session of selected osteopathic diaphragmatic techniques are able to affect muscle motility and thickness, assessed by ultrasounds, in a sample of healthy subjects and to compare results versus a group receiving a sham therapy and another one of non-treated subjects.

DETAILED DESCRIPTION:
Introduction The diaphragm is the dome-shaped sheet of muscle and tendon that serves as the main muscle of respiration and plays a vital role in the breathing process. Also known as the thoracic diaphragm, it represents an important anatomical landmark that separates the chest, from the abdomen.

Indeed, the diaphragm muscle extends from the trigeminal system to the pelvic floor, passing from the thoracic diaphragm to the floor of the mouth. Apart of its anatomy and related anatomical connections, the abdominal diaphragm has been proved to develop many other pivotal relationships: neurologic, vascular and lymphatic, fascial connections The complex anatomic and bio-mechanic structure of thoracic diaphragm, as well as its widespread influences and interactions with both contiguous and more distant areas of the human body, provide a robust rationale for an osteopathic and manipulative approach.

Traditional osteopathy, as presented by the Canadian College of Osteopathy, is defined as: "A natural medicine which aims to restore function in the body by treating the causes of pain and imbalance. To achieve this goal the Osteopathic Manual Practitioner relies on the quality and finesse of his/her palpation and works with the position, mobility and quality of the tissues." A wide number of osteopathic techniques focusing on diaphragm have been proposed but, although systematically and efficiently used, there is a general lack of evidences able to clarify how and to which extent osteopathic manipulative treatment (OMT) on diaphragm is effective and determines a modification in muscles contractility and motion as well as an objective determination of the benefit on the patients receiving treatment.

In a recent study da Silva and colleagues compared manometry pressures of the lower esophageal sphincter before and immediately after osteopathic intervention in the diaphragm of subject with gastroesophageal reflux founding a positive increase in the pressures soon after osteopathic treatment ; however, the estimation of the impact of OMT on diaphragmatic activity was indirect and did not provide any information about changes in motility and contractility; in another large double-blinded, randomized, controlled trial, four hundred and six hospitalized subjects with pneumonia were randomized to receive conventional care only, light touch treatment or OMT, including the doming technique of the diaphragm, in adjunction to conventional treatment for pneumonia. Authors found a significantly shorter length of stay in the OMT and light touch groups vs controls but, once again, they were not able to provide any causal relationship between OMT and diaphragmatic activity . Finally, the effect of OMT in COPD patients has been investigated with contrasting results: in a study on 35 subjects OMT protocol consisted of seven standardized osteopathic manipulative techniques including indirect myofascial re-doming of the diaphragm was compared with sham therapy. Interestingly, results suggest an overall worsening of air trapping during the 30 minutes immediately following one multi - technique OMT session relative to the sham group . Under an indirect point of view, this result favors a role of OMT in diaphragm mobility reactivation, since it may be related to a dynamic hyperinflation-like mechanism promoting air trapping. On the other side another study demonstrated an improved lung function in severely obstructed subjects with COPD following OMT. Thanks to the new hand-held ultrasound instruments, the morphology and function of the diaphragm can be assessed in different settings, such as outpatient clinic, pulmonary function test laboratory, hospital department and intensive care unit, and under different conditions. Ultrasonography is the only non-invasive, non-ionizing imaging technique widely available to directly assess diaphragmatic function. Two different sonographic approaches permit the assessment of muscle thickening in the zone of apposition and excursion of the dome of the diaphragm.

This study therefore aims at investigating whether, to which extent, and how, a single session of selected osteopathic diaphragmatic techniques is able to affect muscle motility and thickness, assessed by ultrasounds, in a sample of healthy subjects and to compare results versus a group receiving a sham therapy and another one of non-treated subjects.

Materials and Methods:

A prospective, randomized, double blinded case vs sham vs control designed study will be conducted.

Seventy-one healthy volunteers will be selected after obtaining written informed consent . A comprehensive clinical history will be obtained in order to identify active or relevant conditions included in the exclusion criteria list.

The remaining participants will be randomized into three arms (experimental, sham therapy and control).

The choice of recruiting healthy volunteers was oriented by the current lack of clear and objective evidences on the impact of osteopathic techniques on the thoraco-abdominal diaphragm. Therefore, since we were not aware of the potential influence of the osteopathic treatment on diaphragmatic motion and function, we judged the identification of a diseased population suitable for treatment an arbitrary choice and excluded subjects with known, proved, or likely diaphragmatic dysfunction.

Study design: all participants, regardless of the assigned group, will receive a comprehensive ultrasonographic evaluation of diaphragmatic motion and thickness (see further) followed by a systematic osteopathic evaluation of the diaphragm. Following, subjects underwent a differential intervention according to their belonging study group: the control group will be simply observed while lying down over the operator's table without receiving any treatment, the shame therapy group will receive a light touch approach (a gently pressure over the chest and subcostal area without any therapeutic purpose) while the experimental group will be effectively treated . After that, a new osteopathic evaluation, followed by a repeated ultrasonography, will be performed in all subjects.

Noteworthy, the study will provide a double blinded design with both, the patient and the ultrasonographist, unaware of the randomization group. Furthermore, the osteopath operator will have no access to the ultrasounds measurement and won't be influenced by it.

Osteopathic evaluation The techniques used to osteopathically assess the diaphragmatic function have been discussed more in details elsewhere.

Ultrasound Evaluation Three consecutive M-mode and Bi-mode measurements of right diaphragm motion will be systematically obtained. A subcostal scan by using a convex probe and frequencies between 2.5 and 3.5 mHz will be achieved during subject's deep inspiration (inspiratory reserve capacity), starting from functional residual capacity, according to described protocols. After that, three estimations of the diaphragmatic strength by measuring diaphragm thickness at end inspiration and end-expiration will be obtained with a longitudinal scan using a linear probe at 12 mHz frequencies. The highest of the three obtained values will finally be collected.

Data Analysis Pre and post osteopathic treatment ultrasound evaluations will be compared in order to detect statistically significant differences in motion and thickness. Secondary aims will be to find out whether clinical, demography or lifestyle factors may be predictors of response to treatment. Finally, the correlation between manual osteopathic assessment and ultrasound measurements will be searched.

ELIGIBILITY:
Inclusion Criteria:

* age below 18 years old

Exclusion Criteria:

* Any current or previous disease, pharmacological treatment or condition contraindicating the manual approach.
* Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessing the change in diaphragm mobility induced by osteopathic treatment | 15 min

SECONDARY OUTCOMES:
Assessing the correlation between osteopathic manual evaluation of diaphragmatic motion and ultrasound measures of mobility | 15 min

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bordoni B, Zanier E. Anatomic connections of the diaphragm: influence of respiration on the body system. J Multidiscip Healthc. 2013 Jul 25;6:281-91. doi: 10.2147/JMDH.S45443. Print 2013. PMID 23940419
- [Background] da Silva RC, de Sa CC, Pascual-Vaca AO, de Souza Fontes LH, Herbella Fernandes FA, Dib RA, Blanco CR, Queiroz RA, Navarro-Rodriguez T. Increase of lower esophageal sphincter pressure after osteopathic intervention on the diaphragm in patients with gastroesophageal reflux. Dis Esophagus. 2013 Jul;26(5):451-6. doi: 10.1111/j.1442-2050.2012.01372.x. Epub 2012 Jun 7. PMID 22676647
- [Background] Noll DR, Degenhardt BF, Morley TF, Blais FX, Hortos KA, Hensel K, Johnson JC, Pasta DJ, Stoll ST. Efficacy of osteopathic manipulation as an adjunctive treatment for hospitalized patients with pneumonia: a randomized controlled trial. Osteopath Med Prim Care. 2010 Mar 19;4:2. doi: 10.1186/1750-4732-4-2. PMID 20302619
- [Background] Noll DR, Degenhardt BF, Johnson JC, Burt SA. Immediate effects of osteopathic manipulative treatment in elderly patients with chronic obstructive pulmonary disease. J Am Osteopath Assoc. 2008 May;108(5):251-9. PMID 18519835
- [Background] Zanotti E, Berardinelli P, Bizzarri C, Civardi A, Manstretta A, Rossetti S, Fracchia C. Osteopathic manipulative treatment effectiveness in severe chronic obstructive pulmonary disease: a pilot study. Complement Ther Med. 2012 Feb-Apr;20(1-2):16-22. doi: 10.1016/j.ctim.2011.10.008. Epub 2011 Nov 27. PMID 22305244
- [Background] Sferrazza Papa GF, Pellegrino GM, Di Marco F, Imeri G, Brochard L, Goligher E, Centanni S. A Review of the Ultrasound Assessment of Diaphragmatic Function in Clinical Practice. Respiration. 2016;91(5):403-11. doi: 10.1159/000446518. Epub 2016 May 25. PMID 27216909